CLINICAL TRIAL: NCT04862858
Title: Improving Outcomes in Patients With Comorbid T2DM and ASCVD: Population Health Management Interventions Supporting Guideline-recommended SGLT2i and GLP-1 RA Medications
Brief Title: Educational Intervention to Increase Select Guideline-recommended Cardioprotective Medications in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Humana Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry); Humana Healthcare Research, Inc. (Unknown)
Responsible Party: Principal Investigator, Alexjandro Daviano, Research Consulting Lead, Humana Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1236
Record Dates: First submitted 2021-04-12; First posted 2021-04-28 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The educational outreach intervention will entail a multi-faced strategy to provide patients resources to learn more about reducing their risk for heart disease and supporting providers in the care of their patients by sharing recent guideline-recommended treatments for these high-risk individuals.
  Interventions: Other: Educational Intervention
- Control (No Intervention): Patients and primary care providers randomly selected and assigned to the control arm will not receive any of the educational outreach communications.

INTERVENTIONS:
Other: Educational Intervention — The educational intervention will involve guideline-based treatment recommendation information for providers via fax/mail and phone and provide resources via mail and phone for patients to learn more about ways to reduce their cardiovascular risk.
  Arms: Intervention

SUMMARY:
This is an educational outreach to patients with type 2 diabetes mellitus (T2DM) and atherosclerotic cardiovascular disease (ASCVD) and their primary care and specialist providers to improve use of guideline-recommended treatments, specifically sodium-glucose cotransporter 2 inhibitor (SGLT2i) and glucagon-like peptide-1 receptor agonist (GLP-1 RA) medications.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus, a history of atherosclerotic cardiovascular disease, without use of select guideline-recommended medications in the previous year will be identified from administrative claims. Primary care providers will be identified, randomly selected and randomized to the intervention arm or control arm. All eligible patients for that provider will be included. The patient's specialist providers (cardiologist and/or endocrinologist, as applicable) will be identified and contacted. The intervention will include a multi-faceted strategy to support providers in the care of their patients by sharing recent guideline-based treatment recommendations and provide patients with information regarding ways to reduce their cardiovascular risk. Outreach will occur for all patients and providers randomized for the intervention - there will be no active enrollment or recruitment.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Patients with T2DM defined as ≥2 outpatient diagnoses of T2DM in any position on separate days; OR ≥1 inpatient diagnosis T2DM in any position; OR ≥1 outpatient diagnosis in any position AND ≥1 medication claim for T2DM
* ≥1 diagnosis code for ASCVD (coronary artery disease diagnoses or procedures, cerebrovascular disease, peripheral artery disease of atherosclerotic origin) on any claim type in any position within the 24-month period prior to identification
* Enrolled in a Humana Medicare Advantage Prescription Drug plan with ≥12 months pre-identification continuous enrollment (no more than a 31 day gap) as of the identification date and currently enrolled as of the identification date
* Age 18-85 years at time of identification
* Patients residing in Kentucky (KY), West Virginia (WV), Pennsylvania (PA), and 6 counties in south New Jersey (NJ) (Burlington, Camden, Cumberland, Gloucester, Mercer, Salem) (United States)

Provider

* Primary care providers of the identified patients

Exclusion Criteria:

Patients

* ≥1 diagnosis or procedure code for end-stage kidney disease, renal transplant, dialysis or kidney failure
* Any hospice or long-term care residence
* ≥1 code for pregnancy/childbirth
* Patients with any use of SGLT2i or GLP-1 RA medications in the pre-identification period
* Patients without an attributed primary care provider
* Patients on do not contact lists
* Patients without valid addresses and telephone numbers
* Patients with ≥1 diagnosis for type 1 diabetes pre-identification

Primary care providers

* Providers on do not contact lists
* Providers without valid fax/mailing address and phone number
* Providers with <3 or >50 eligible patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4197 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-08-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of individuals who initiate guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, based on administrative claims data | 6-months
  Percentage of individuals with T2D & ASCVD who have ≥1 pharmacy claim for SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products

SECONDARY OUTCOMES:
Percentage of individuals who initiate guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, based on administrative claims data | 12-months
  Percentage of individuals with T2D & ASCVD who have ≥1 pharmacy claim for SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products
Percentage of individuals adherent to guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, based on administrative claims data | 6-months
  Adherence to guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, measured by proportion of days covered based on days' supply of medications from pharmacy claims
Percentage of individuals persistent to guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, based on administrative claims data | 6-months
  Persistence to guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, excluding combination products, measured by <90 day gap in treatment based on pharmacy claims
Percentage of individuals who initiate guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, including combination products, based on administrative claims data | 6-months
  Percentage of individuals with T2D & ASCVD who have ≥1 pharmacy claim for SGLT2i or GLP-1 RA medications with cardiovascular benefit, including combination products
Percentage of individuals who initiate guideline-based SGLT2i or GLP-1 RA medications with cardiovascular benefit, including combination products, based on administrative claims data | 12-months
  Percentage of individuals with T2D & ASCVD who have ≥1 pharmacy claim for SGLT2i or GLP-1 RA medications with cardiovascular benefit, including combination products

CONTACTS AND LOCATIONS:
Overall Officials: Alexjandro Daviano, DN, DrPH, Principal Investigator — Humana Inc.
Locations (1):
- Humana, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S111-S124. doi: 10.2337/dc21-S009. PMID 33298420
- [Background] American Diabetes Association. 10. Cardiovascular Disease and Risk Management: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S125-S150. doi: 10.2337/dc21-S010. PMID 33298421
- [Background] Das SR, Everett BM, Birtcher KK, Brown JM, Januzzi JL Jr, Kalyani RR, Kosiborod M, Magwire M, Morris PB, Neumiller JJ, Sperling LS. 2020 Expert Consensus Decision Pathway on Novel Therapies for Cardiovascular Risk Reduction in Patients With Type 2 Diabetes: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2020 Sep 1;76(9):1117-1145. doi: 10.1016/j.jacc.2020.05.037. Epub 2020 Aug 5. No abstract available. PMID 32771263

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT04862858/Prot_SAP_000.pdf